CLINICAL TRIAL: NCT00135967
Title: Treatment of Patients With Membranous Nephropathy and Renal Insufficiency With Mycophenolate Mofetil and Prednisone: a Pilot Study
Brief Title: Mycophenolate Mofetil in Membranous Nephropathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RUNMN02
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2005-12-06 (Estimated); Status verified 2005-08

CONDITIONS: Glomerulonephritis, Membranous
Keywords: membranous nephropathy; mycophenolate mofetil; cyclophosphamide; prednisone
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — BID protein, human; Methylprednisolone

INTERVENTIONS:
Drug: mycophenolate mofetil orally 1000 mg twice a day (BID)
Drug: prednisone 0,5 mg/kg orally on alternate days
Drug: intravenous (i.v.) methylprednisolone 1000 mg, total 9

SUMMARY:
Patients with idiopathic membranous nephropathy and renal insufficiency are at risk for end-stage renal disease (ESRD). Treatment with cyclophosphamide is currently used as a treatment modality. Mycophenolate mofetil is a new immunosuppressive agent with fewer side effects.

In this pilot study patients with membranous nephropathy and renal failure will be treated with mycophenolate mofetil and prednisone. The outcome will be compared with historical controls treated with a similar regimen containing cyclophosphamide.

ELIGIBILITY:
Inclusion Criteria:

* Membranous nephropathy
* Serum creatinine (Screat)> 1,5 mg/dl or ECC < 70 ml/min or increase Screat > 50%
* Proteinuria > 2 g/day

Exclusion Criteria:

* Systemic diseases
* Pregnancy wish
* Active infection
* Liver dysfunction
* Abnormal hematology lab
* Unstable angina
* Nonsteroidal anti-inflammatory agents (NSAIDs)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-05

PRIMARY OUTCOMES:
renal function (serum creatinine)
proteinuria

SECONDARY OUTCOMES:
side effects
relapse rate

CONTACTS AND LOCATIONS:
Overall Officials: Jack F Wetzels, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Department of Nephrology Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Branten AJ, du Buf-Vereijken PW, Vervloet M, Wetzels JF. Mycophenolate mofetil in idiopathic membranous nephropathy: a clinical trial with comparison to a historic control group treated with cyclophosphamide. Am J Kidney Dis. 2007 Aug;50(2):248-56. doi: 10.1053/j.ajkd.2007.05.015. PMID 17660026